CLINICAL TRIAL: NCT00845572
Title: The Consta Club: A Demonstration Project for Setting up a Consta Club in a Community Mental Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20070020H
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia; Schizoaffective
Keywords: Schizophrenia; Schizoaffective; Risperdal Consta; Medication Adherence; Antipsychotic
MeSH Terms: conditions — Schizophrenia; Medication Adherence | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Consta Club (Experimental)
  Interventions: Behavioral: Consta Club

INTERVENTIONS:
Behavioral: Consta Club — Biweekly group for patients receiving Risperdal Consta injections. Each 45 minute group includes socialization time, goal-setting, illness and medication education, and refreshments.
  Other Names: Risperdal Consta

SUMMARY:
This study will establish a bi-weekly Consta Club. Participants will begin taking Risperdal Consta after being recommended by their treating physician. As a part of the Consta Club attendees will receive their injection of Risperdal Consta and be educated about important mental health issues. Interviews with study participants will be completed every three months to determine the effectiveness of the change to Risperdal Consta and the bi-weekly group. The overall hypothesis is that the individuals in Consta Club will have a decrease in walk-in visits, emergency procedures and hospitalizations. It is also believed that individuals in Consta Club will have fewer symptoms and better levels of functioning.

DETAILED DESCRIPTION:
Poor adherence to oral antipsychotic medication leads to rehospitalization, derails the process of recovery, and contributes to the high cost of treating schizophrenia. Unfortunately, poor adherence is common for individuals with this diagnosis. An organizing hypothesis of our research program is that forgetfulness and failure to establish a routine that facilitates medication adherence are prominent reasons for non-adherence.

We have established a thirty minute bi-weekly Consta Club in which individuals will attend a social group and and also receive their injection of Risperdal Consta. Consta Club will educate individuals about the importance of medication adherence as well as establish a routine that facilitates adherence. The club will provide the opportunity for the club members to discuss their mental illness, develop goals to recovery, establish a means of transportation to the club and participate in drawings to win prizes. The overall hypothesis is that the individuals in Consta Club will experience a decrease in walk-in visits, emergency procedures and hospitalizations. It is also hypothesized that individuals in Consta Club will demonstrate lower levels of symptomatology, higher levels of quality of life and improvements in functioning when compared to their baseline.

A total of twenty-five individuals will be recruited to switch from an oral atypical antipsychotic medication to Risperdal Consta which will be supplied by Janssen Pharmaceutica at no cost to the individual or the clinic. Individuals will be recruited prior to hospital discharge if inpatient at time of recruitment OR from the local mental health clinic. Hospitalized individuals will be started on Risperdal Consta prior to discharge and outpatients will switch from oral atypical antipsychotics within two weeks. Individuals will be receiving a single injection of Risperdal Consta every two weeks. Prior to the switch and every 3 months for a period of 9 months the individual will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are able to understand the consent form and who have given informed consent.
2. Between the ages of 18 and 65.
3. Diagnosis of schizophrenia or schizoaffective disorder
4. Receiving treatment with an oral atypical antipsychotic medication for at least two months prior to study
5. Only partial adherence (80% or less) to antipsychotic medication
6. If they have tried Consta but did not receive an adequate trial and did not experience any adverse symptoms.
7. Some responsibility for attending Consta Club meetings and injections.
8. Able to understand and complete rating scales.

Exclusion Criteria:

1. History of significant head trauma, seizure disorder, or mental retardation.
2. Has a legal guardian.
3. Alcohol or drug abuse or dependence within the past 3 months.
4. Previous negative reactions to oral Risperdal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Service Utilization - Patients in consta club will have fewer missed visits, fewer unscheduled visits, and fewer emergency visits and hospitalizations than matched patients on oral antipsychotics | end of study

SECONDARY OUTCOMES:
Patients in consta club will demonstrate lower levels of symptomatology and higher levels of quality of life and community adjustment than matched patients on oral antipsychotics | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Dawn' I Velligan, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States